CLINICAL TRIAL: NCT03860051
Title: Association Between Lactase Deficiency, Symptoms of Lactose Intolerance, and the Small Intestinal Microbiome in Adults
Brief Title: Association Between Lactase Deficiency, and the Small Intestinal Microbiome in Adults.
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Huiping Xu, Associate Professor, Indiana University
Other Study IDs: 1805571295
Record Dates: First submitted 2019-02-27; First posted 2019-03-01 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Lactose Intolerance
MeSH Terms: conditions — Lactose Intolerance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Endoscopy and Biopsy Sampling:
  Four post-bulbar mucosal biopsy samples will be taken using standard biopsy forceps from each patient. Two biopsy samples will be placed in a small, tightly capped plastic tube without any supporting media. Two biopsy samples will be submerged in Allprotect ® Tissue Reagent (Qiagen) for immediate stabilization of DNA, RNA, and protein and archived at -20 to -80 degrees Celsius for long-term storage for planned small bowel microbiome analyses.
  Fecal Microbiome:
  Stool samples will be collected and archived at -80 degrees Celsius for future analysis of the fecal microbiome
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to study the role of the enzyme (substance produced by the body that helps in a biochemical reaction like digestion in the body) responsible for digestion of lactose and the role of the gut bacteria (bacteria in the intestine) in producing symptoms of lactose intolerance.

DETAILED DESCRIPTION:
The study involves 3 visits and will include 2 types of subjects - those who have the the diagnosis of lactose intolerance (subjects) and those who do not have lactose intolerance (controls).

Visit 1:

In total, it is estimated that the research participation will add about 1 hour to your planned procedure visit. At Visit 1 following will be done

* Subjects will be asked to read and sign the informed consent after all the questions about the study have been answered.
* General medical history will be taken including demographics, symptoms and history of illness, and medication review.
* Vital signs (blood pressure, temperature, respiration, height, and weight) will be recorded.
* Subjects will be asked to complete 2 questionnaires
* Upper endoscopy will be done as part of routine clinical care
* At the time of the endoscopy 4 extra biopsies (small piece of tissue) from the small intestines will be taken. The biopsies will be used for research to detect the bacteria and to measure the lactase enzyme.
* Small sample of blood (10 mL) (2 teaspoons) will be taken for storage for possible future testing. This will be a one time draw only.
* The research team may contact the subjects to arrange a Visit 2 if they are interested in proceeding with the next step in this research study.

Visit 2:

Visit 2 will take approximately 6 hours to complete. If the subject returns for Visit 2, they will do the following

* They will return to the research office at Indiana University to participate in hydrogen breath test (test that uses the measurement of hydrogen in the breath to diagnose several conditions) to see how the body reacts to lactose. This involves drinking milk, then blowing into a bag so we can collect breath samples. Subjects will be asked to report any symptoms they might have during this time. This test will take approximately 6 hours. They will be instructed to eat a low-fiber meal the night before the test, and asked to fast for the 12 hours before the test. They can drink water during this time.
* They will be also be asked to provide a stool sample for future analysis. Instructions for collection, storage and transportation of stool will be provided. They will be provided a kit for stool collection, storage and transportation. They will be asked to collect stool at home over the course of 2 days and store as per instructions. Stool will need to be refrigerated and brought back to the office on ice.

Visit 3:

Visit 3 will take approximately less than one hour to complete. For those who are interested in returning for Visit 3,

* Subjects will be asked to return to the clinic with the stool samples.
* They will complete the study at this time.

Participants who complete Aim 1 and meet further eligibility criteria for Aim 2 may be contacted by research staff to return for Visit 2 (breath test). Those who are agreeable to participating and are scheduled for Visit 2 will be instructed to consume a low-fiber meal and fast for 12 hours prior to their breath test. We will contact the participant 24 to 48 hours prior to the test day as a reminder to consume a low fiber meal and fast for 12 hours.

ELIGIBILITY:
Patient ages 18-75 presenting for upper gastrointestinal endoscopy for any indication except those outlined in the exclusion criteria below at the IU GI Endoscopy Sites including: IU North Hospital, Glen Lehman Endoscopy Suite, Springmill/Beltway Surgery Center, IU Saxony, and Eskenazi Hospital will be eligible for participation. Participants should be willing and able to sign informed consent.

Inclusion Criteria for Controls (Aim 1): Adult patients ages 18-75 years meeting basic eligibility criteria as listed above will be considered for inclusion. Participants should report no current or recent history of intolerance to and avoidance of dairy nor use of treatments and products for dairy intolerance.

Inclusion Criteria for Patients with Self-Reported Lactose Intolerance (Aim 1): Adult patients ages 18-75 years meeting basic eligibility criteria as listed above will be considered for inclusion. Participants should report current or recent history of intolerance to and avoidance of dairy.

Inclusion Criteria for Controls (Aim 2): All controls eligible for and completing Aim 1 will be considered eligible for inclusion. Participants should not meet any of the Aim 2 exclusion criteria.

Inclusion Criteria for Patients with Self-Reported Lactose Intolerance (Aim 1): All patients with self-reported lactose intolerance eligible for and completing Aim 1 will be considered eligible for inclusion. Participants should not meet any of the Aim 2 exclusion criteria.

Exclusion criteria (Aim 1):

1. Patients with known bleeding diathesis given the need for small intestinal mucosal biopsies.
2. Patients with known history of eosinophilic esophagitis, inflammatory bowel disease, chronic pancreatitis or pancreatic insufficiency, celiac disease, peptic duodenitis
3. Antibiotic-use within the last 30 days
4. Major abdominal surgery except appendectomy or cholecystectomy > 6 months prior to enrollment
5. Prior radiation therapy of the abdomen
6. Use of tobacco products within the last 3 months
7. Allergy to milk
8. Currently pregnant or breast-feeding
9. Patients taking anti-coagulant drugs

Exclusion criteria (Aim 2):

1. Meeting any of the exclusion criteria as listed for Aim 1
2. Known diagnosis of disorders associated with abnormal GI motility (gastroparesis, amyloidosis, neuromuscular disease including Parkinson's disease, collagen vascular disease, chronic malnutrition, and uncontrolled thyroid disease)
3. History of small intestinal bacterial overgrowth
4. Active peptic ulcer disease noted at the time of endoscopy
5. Recent colonoscopy bowel preparation or colonic enema in the preceding 4 weeks
6. Chronic immunodeficiency or chronic infectious illness
7. Currently undergoing chemotherapy
8. Patients taking anti-coagulant drugs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient ages 18-75 presenting for upper gastrointestinal endoscopy for any indication except those outlined in the exclusion criteria below at the IU GI Endoscopy Sites including: IU North Hospital, Glen Lehman Endoscopy Suite, Springmill/Beltway Surgery Center, IU Saxony, and Eskenazi Hospital will be eligible for participation. Participants should be willing and able to sign informed consent.
Sampling Method: Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2018-11-21 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Lactase activity | 1 day
  Lactase activity (µmol/min/g) will be assessed from small bowel biopsy specimens

SECONDARY OUTCOMES:
Symptom severity | 1 day
  We will assess symptom severity using the lactose assessment tool
Small intestinal mucosal microbiome | 1 day
  The small intestinal microbiome will be assessed by 16S allele PCR sequencing (16S) and Shotgun Metagenomic Sequencing (SGS)
Maldigestion status | 1 day
  Maldigestion status will be assessed by hydrogen breath test
Fecal microbiome | 1 day
  The fecal microbiome will be assessed by 16S allele PCR sequencing (16S) and Shotgun Metagenomic Sequencing (SGS)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea S Shin, MD, Principal Investigator — IU
Locations (1):
- Indiana University Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No